CLINICAL TRIAL: NCT04289896
Title: Effectiveness of an Intervention Through a Plyometric Training Program, in the Improvement of Explosive Strength and Speed in Youth Players. A Randomized Clinical Study.
Brief Title: Plyometric Training, in the Improvement of Explosive Strength and Speed in Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PLYO
Record Dates: First submitted 2020-02-27; First posted 2020-02-28 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Football Player
Keywords: Football, Youth players; Plyometric exercises; Strength; Running speed; Muscular extensibility; Youth players
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Each session will last 20 minutes, taking place 2 days a week, for a period of 4 weeks. Prior to the completion of the routine training of each team, the plyometric exercise program will be carried out in the experimental group. When the intervention ends, the members of the experimental group will perform the usual training
  Interventions: Other: Plyometric exercise
- Control group (No Intervention): Athletes included in the control group will not perform any intervention, continuing with their usual routine.

INTERVENTIONS:
Other: Plyometric exercise — The plyometric program to be followed by the subjects assigned to the experimental group during the four weeks includes: Squat jumps, alternate lunge, cyclic horizontal jump, horizontal left leg jump, horizontal right leg jump, vertical left leg jump, right leg vertical jump, squat box jumps, box jumps left leg, box jumps right leg, box to box squat jumps, box to box left leg, box to box right leg.
  In all the exercises the subjects will be able to help themselves with the arms and a rest period of 120 seconds will be left between each series.
  The intervention will be carried out prior to training, keeping a minimum of 48 hours of rest between sessions.
  Arms: Experimental group

SUMMARY:
Football requires a high number of actions at high speed and intensity. The application of plyometrics can improve explosive strength and speed levels in soccer players.

The main objective of the study is to assess the effectiveness of a program based on plyometric exercises for the improvement of the explosive force in vertical jump and the speed in running with and without the ball in soccer players of youth category.

Randomized clinical study, simple blind, with follow-up period. 30 players will be randomized to the study groups: experimental and control. The intervention will last 4 weeks, with 2 weekly sessions lasting 20 minutes. The study variables will be: Vertical Countermovement Jump Test with Arms and Twenty-Centimeter Drop Jump Reactive Strength Index (Explosive Force), running speed without ball and ball (20 meter speed test), hitting speed of ball (Maximal Kicking Velocity Test), hamstring extensibility (Sit and Reach Test) and sural triceps extensibility (Leg Motion Basic). Normality will be calculated using an analysis of Kolmogorov Smirnov. With the t-student test the differences between assessments will be calculated and with an ANOVA of repeated measures, the effect between intersubject will be calculated. The effect size will be obtained with Cohen's formula.

It is expected to obtain an improvement in the explosive force in the vertical jump, as well as in the running speed with and without the ball.

ELIGIBILITY:
Inclusion Criteria:

* Youth soccer players federated in Castilla y León
* Over 18 years
* Male
* That they train at least twice a week.

Exclusion Criteria:

* subjects who: present a medical diagnosis of musculoskeletal lesion in the lower limb at the time of starting the study
* Who have been out of the competition for more than 6 months as a result of an injury in the last year
* That are part of the experimental phase of another study during our intervention and follow-up period
* That they do not attend at least 80% of the intervention sessions
* Not sign the informed consent document.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline explosive force in vertical jump after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  Through the Vertical Countermovement Jump Test with Arms. The subject will be placed in standing position on a contact platform, it should make a rapid downward movement followed by a maximum vertical jump using the arms. The distance jumped in centimeters will be measured.

SECONDARY OUTCOMES:
Change from baseline running speed after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  A speed test of 20 meters will be carried out on a flat surface of grass, which will be carried out both with a ball and without a ball. Initially, there will be a specific warm-up of 3 sub-maximum races in those 20 meters, after which, the subjects will make 3 maximum sprints of 20 meters, with 3 minutes of rest between them. The race will start with the subject 0.5 meters behind the starting line. The time it takes for the subject to arrive from the start line to the 20 meter line will be measured. The fastest sprint time of the 3 attempts will be selected.
Change from baseline ball hitting speed after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  Through the Maximal Kicking Velocity Test. Each subject will hit a soccer ball located on the ground, instructing them to obtain maximum speed. They must strike with maximum force towards a net with the dominant leg and with a run of 2 strides. The distance between the ball and the net will be 4 meters. Each subject will make 2 practice strokes and 3 strokes of maximum strength, among which 1 minute rest will be allowed. The speed of the ball will be measured with a radar placed 2 meters from the ball and 0.7 meters from the ground
Change from baseline hamstring extensibility after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  It will be done by applying the Sit and Reach Test. This test will be carried out with the subject seated, knees extended and the feet in 90º of flexion placed both, against a drawer designed for the realization of this test. From this position, the subject is urged to progressively and maximally flex the trunk with the legs and arms extended while maintaining the final position for 2 seconds. The final position is the result of the test, assessing at that time the distance (in centimeters) that exists between the tips of the fingers and the tangent to the soles of the feet
Change from baseline sural triceps extensibility after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  An assessment of the dorsiflexion of the ankle under load will be performed. It will be used as a measuring instrument Leg Motion Basic. The subject will be placed in standing position (arms crossed on the chest) with the foot to be assessed in advance on the work surface, respecting the marks of this. You should perform an ankle dorsiflexion forward the knee while moving the vertical reference on the platform. It is important to ensure that the subject does not detach the heel from the floor during the test

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain